CLINICAL TRIAL: NCT01310361
Title: Once-daily Therapy for Streptococcal Pharyngitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Azad University of Medical Sciences (Other)
Responsible Party: Reasercheal Deputy of Islamic Azad University ,Mashhad Branch,Mashhad,Iran., Islamic Azad University ,Mashhad Branch,Mashhad,Iran.
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: iaum
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2005-01

CONDITIONS: Streptococcal Sore Throat
Keywords: Pharyngitis; Group A β-hemolytic Streptococci; Exudate; Erythema Penicillin; Amoxicillin
MeSH Terms: conditions — Pharyngitis | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amoxicillin (Experimental): Once-daily Therapy for Streptococcal Pharyngitis With Amoxicillin
  Interventions: Drug: Amoxicillin
- Benzathin Penicillin G (Active Comparator): Once-daily Therapy for Streptococcal Pharyngitis With Intramuscular Benzathin Penicillin G
  Interventions: Drug: Intramuscular Benzathin Penicillin G

INTERVENTIONS:
Drug: Amoxicillin
  Arms: Amoxicillin
Drug: Intramuscular Benzathin Penicillin G — It is mentioned underlined in page 10 in research. (Once the throat swab was taken and cultured on plate at the place where the child was examined, hygiene teacher was trained about how to prepare the oral amoxicillin suspension and how to give it to the child. 750 milligrams of amoxicillin was thereafter given to the patient and in order not to infect other school children, the patient was sent home. The following morning, the patient would come to school and was given the second dose of amoxicillin by the hygiene teacher. All oral drugs were bought from a creditable company. In the injection group, 600000 units of penicillin was administered to children who weigh less than 27 kilograms and 1200000 units of penicillin was administered to children who weigh more. After 48 hours, patients were examined again when the result of first culture was ready)
  Arms: Benzathin Penicillin G

SUMMARY:
In some studies once daily amoxicillin therapy might be treatment of choice for Group A β-hemolytic Streptococcus pharyngitis in comparison with three to four times daily treatment with oral penicillin V.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

1. Age of 6 to 15 years old.
2. The criteria in clinical examination including objective signs (fever, Erythema or exudate of tonsils, enlarged lymph nodes) and subjective sign(sore throat). Neck tenderness, abdominal pain and pharynx petechia were also considered.
3. No antibiotic was used during the week before.
4. -Performing throat culture before the initiation of drug administration
5. Positive throat culture indication GABHS
6. No previous history of allergy to penicillin .

Exclusion Criteria:

1. Age of below 6 years old or above 15 years old.
2. No signs of pharyngitis in the clinical examination
3. Antibiotic use during the week before.
4. Throat culture was not performed before the initiation of drug administration.
5. Negative throat culture or the culture indicates a microorganism other than GABHS.
6. History of allergy to penicillin
7. Not using drugs or not following the treatment in the field of having the second culture performed.

Ages: 6 Years to 15 Years | Sex: All
Age Groups: Child
Dates: Start 2004-01; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Locations (1):
- Islamic Azad University, Mashhad, Khorasan, Iran